CLINICAL TRIAL: NCT01168505
Title: The Role of Intravenous Iron to Prevent Anemia in Women With Breast Cancer Receiving (Neo)Adjuvant Chemotherapy
Brief Title: Iron Supplement in the Prevention of Anemia in Female Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Fundação Faculdade de Medicina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NP 002/2009 - CEP 543/09
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — teferrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- no iron supplentation (No Intervention)
- iron supplement (Experimental)
  Interventions: Drug: ferric hydroxide saccharate

INTERVENTIONS:
Drug: ferric hydroxide saccharate — single dose of 200 mg (2 ampoules), 24-48 hours after administration of chemotherapy for a total of four doses
  Other Names: NORIPURUM
  Arms: iron supplement

SUMMARY:
Study to evaluate the efficacy of intravenous iron supplementation in the prevention of anemia in patients receiving (neo)adjuvant breast cancer regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Women older than 18 years
2. Patient with operated breast cancer with indication for (NEO)adjuvant therapy
3. They must have hemoglobin levels within the normal range (> 12g/dL), absence of renal and hepatic dysfunction as assessed by serum levels of urea, creatinine, AST, ALT.
4. Lack of folic acid deficiency and vitamin B12
5. Able to provide written informed consent.

Exclusion Criteria:

1. Use of any oral supplement containing iron;
2. Patients who have iron overload as defined by serum ferritin> 800 microg / L or transferrin saturation> 40%;
3. Patients who are pregnant or breastfeeding;
4. History of active infection or active bleeding except menstruation;
5. History of HIV or hepatitis B or C - clinically important; -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of intravenous iron supplementation in the prevention of anemia in patients receiving (neo)adjuvant breast cancer regimens | 18 weeks
  Anemia prevention defined by hemoglobin levels

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Hoff, MD Professor, Principal Investigator — Instituto do Câncer do Estado de São Paulo
Locations (2):
- Brazil (2):
  - Instituto Do Cancer Do Estado de São Paulo, São Paulo, São Paulo
  - Hospital Sirio Libanes, São Paulo, São Paulo